CLINICAL TRIAL: NCT05498701
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, CROSSOVER, SINGLE DOSE STUDY TO DETERMINE THE BIOEQUIVALENCE OF 12.2 MG TAFAMIDIS FREE ACID TABLETS AND COMMERCIAL 20 MG TAFAMIDIS MEGLUMINE CAPSULES ADMINISTERED UNDER FASTED CONDITIONS AND THE EFFECT OF FOOD ON ORAL BIOAVAILABILITY OF 12.2 MG TAFAMIDIS FREE ACID TABLETS IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study Comparing Two Forms of Tafamidis Without Food and the Amount of Tafamidis in the Blood With Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461103
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Tafamidis, B3461103
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test tablet (fasted) followed by Reference capsule (fasted) followed by Test tablet (fed) (Experimental): On Day 1 of each period, participants will receive a single dose of one of the tafamidis formulations under fasted or fed conditions. Each period is separated by a washout of at least 16 days between administration of study drug.
  Interventions: Drug: Tafamidis free acid tablet (Test); Drug: Tafamidis meglumine capsule (Reference)
- Reference capsule (fasted) followed by Test tablet (fasted) followed by Test tablet (fed) (Experimental): On Day 1 of each period, participants will receive a single dose of one of the tafamidis formulations under fasted or fed conditions. Each period is separated by a washout of at least 16 days between administration of study drug.
  Interventions: Drug: Tafamidis free acid tablet (Test); Drug: Tafamidis meglumine capsule (Reference)

INTERVENTIONS:
Drug: Tafamidis free acid tablet (Test) — 12.2 mg tafamidis free acid tablet (Test)
Drug: Tafamidis meglumine capsule (Reference) — Commercial 20 mg tafamidis meglumine capsule (Reference)

SUMMARY:
The purpose of this clinical trial is to compare a tablet and a capsule form of tafamidis without food and to assess the amount of tafamidis in blood after taking the tablet form with food.

This study is seeking healthy participants over the age of 18.

All participants in the study will receive either one tablet or capsule of study medicine on the first day without food, then receive one dose of the other tablet or capsule form 16 days later without food. All participants will then receive one dose of the tablet form with food 16 days later.

We will evaluate the amounts in blood for 8 days after taking each dose of the study medicine.

Participants will take part in this study for about 96 days. The first visit is a screening visit to ensure that participants are appropriate for the study. Up to 28 days later, eligible participants will visit the study clinic three times (and stay overnight in the clinical research center for 8 nights each time). The study team will also call participants over the phone 28 to 35 days after the last dose of medicine.

ELIGIBILITY:
Inclusion Criteria

1. Participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening.
2. Healthy female participants of nonchildbearing potential and/or male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
3. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

Medical Conditions:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
   * Hypersensitivity to any component of the formulations
2. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
3. Use of prescription or nonprescription drugs, dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention. (Refer to Section 6.9 Prior and Concomitant Therapy for additional details).
4. Current use of any prohibited concomitant medication(s) or participant unwilling/unable to use a permitted concomitant medication(s). Refer to Section 6.9 Prior and Concomitant Therapy.

   Prior/Concurrent Clinical Study Experience:
5. Previous administration with an investigational product (drug or vaccine) within 6 months (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

   Diagnostic Assessments:
6. A positive urine drug test.
7. Screening seated BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of seated rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is >450 ms, this interval should be rate-corrected using the Fridericia method only and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * AST or ALT level ≥ 1.5 × ULN;
   * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.

   Other Exclusion Criteria:
10. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
12. History of sensitivity to heparin or heparin induced thrombocytopenia.
13. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
14. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
15. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pharma Medica Research Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 22 participants were enrolled in this study. Eleven participants were randomized to Sequence 1 and 11 participants were randomized to Sequence 2, all 22 participants received study interventions.
Groups:
- Sequence 1: Participants randomized to Sequence 1 received tafamidis free acid tablet 12.2 mg, fasted (Test) in Period 1 followed by commercial tafamidis meglumine soft gelatin capsule 20 mg fasted (Reference) in Period 2 and tafamidis free acid tablet 12.2 mg, fed in Period 3. Each period was separated by a washout of at least 16 days between administration of study drug.
- Sequence 2: Participants randomized to Sequence 2 received commercial tafamidis meglumine soft gelatin capsule 20 mg, fasted (Reference) in Period 1 followed by tafamidis free acid tablet 12.2 mg, fasted (Test) in Period 2 and tafamidis free acid tablet 12.2 mg, fed in Period 3. Each period was separated by a washout of at least 16 days between administration of study drug.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Median (Full Range); unit: Years] | 40.0 [24 to 59] | 37.0 [23 to 67] | 39.5 [23 to 67]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18-25 years | 1 | 2 | 3
  26-35 years | 2 | 3 | 5
  36-45 years | 3 | 2 | 5
  >45 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics(PK) Parameter - Area Under the Concentration-time Curve to Infinity (AUCinf) of PF-06291826
Description: AUCinf is defined as area under the concentration-time curve from time 0 to infinity, and calculated by AUC(0-tlast) + (Clast*/kel), where Clast* is the estimated plasma concentration at the last quantifiable time point (Clast) estimated form the log-linear regression analysis Clast* = Clast x e^(-kel x tlast)
Time Frame: Predose and 0.5, 1,2,3,4,6,8,12,24 (Day 2),48 (Day 3),72 (Day 4),96 (Day 5),120 (Day 6),144 (Day 7), and 168 (Day 8) hours post dose
Population: All participants who received at least 1 dose of tafamidis and who had at least 1 of the PK parameters of interest calculated. Here "Number of Participants Analyzed" signifies participants who contributing to this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms * hour per milliliter
Groups:
- Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted): Participants received a single tafamidis free acid tablet 12.2 mg under fasted condition orally on Day 1 of Period 1 for participants randomized in Sequence 1 and on Day 1 of Period 2 for participants randomized in Sequence 2.
- Tafamidis Meglumine 20 mg Oral Capsule (Fasted): Participants received a single commercial tafamidis meglumine capsule 20 mg orally under fasted condition on Day 1 of Period 2 for participants randomized in Sequence 1 and on Day 1 of Period 1 for participants randomized in Sequence 2.
- Tafamidis Free Acid 12.2 mg Oral Tablet (Fed): Participants received a single tafamidis free acid tablet 12.2 mg orally under fed condition on Day 1 of Period 3 for participants randomized in Sequence 1 and Sequence 2.
Arm/Group | Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) | Tafamidis Meglumine 20 mg Oral Capsule (Fasted) | Tafamidis Free Acid 12.2 mg Oral Tablet (Fed)
Number analyzed (Participants) | 16 | 18 | 17
Nanograms * hour per milliliter | 60670 (24) | 67690 (22) | 60210 (28)
Statistical Analysis 1: Comparison: Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) vs Tafamidis Meglumine 20 mg Oral Capsule (Fasted); Bioequivalence of the Test treatment (Tafamidis free acid 12.2 mg oral tablet [Fasted]) to Reference treatment (Tafamidis meglumine 20 mg oral capsule [Fasted]) was concluded if the 90% confidence intervals for the ratios of adjusted geometric means for tafamidis AUCinf fell entirely within the acceptance region of (80%,125%); Test type: Other; Ratios of Adjusted Geometric Means = 93.19, 90% CI 2-sided [87.10 to 99.70]

2. Primary Outcome: PK Parameter - Maximum Observed Concentration (Cmax) of PF-06291826
Description: Cmax is defined as maximum observed concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) | Tafamidis Meglumine 20 mg Oral Capsule (Fasted) | Tafamidis Free Acid 12.2 mg Oral Tablet (Fed)
Number analyzed (Participants) | 16 | 18 | 17
Nanograms per milliliter | 1046 (19) | 1291 (21) | 891.2 (18)
Statistical Analysis 1: Comparison: Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) vs Tafamidis Meglumine 20 mg Oral Capsule (Fasted); Bioequivalence of the Test treatment (Tafamidis free acid 12.2 mg oral tablet [Fasted]) to Reference treatment (Tafamidis meglumine 20 mg oral capsule [Fasted]) was concluded if the 90% confidence intervals for the ratios of adjusted geometric means for tafamidis Cmax fell entirely within the acceptance region of (80%,125%); Test type: Other; Ratio of Adjusted Geometric Means = 81.00, 90% CI [76.25 to 86.04]

ADVERSE EVENTS:
Time Frame: The time period for collecting AEs for each participant begins from the time the participant provided informed consent up to 35 days after administration of the final dose of study intervention (approximately 11 weeks).
Description: Same event may appear as both a NSAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) | Tafamidis Meglumine 20 mg Oral Capsule (Fasted) | Tafamidis Free Acid 12.2 mg Oral Tablet (Fed)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 4/22 | 2/22 | 4/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tafamidis Free Acid 12.2 mg Oral Tablet (Fasted) (N=22) | Tafamidis Meglumine 20 mg Oral Capsule (Fasted) (N=22) | Tafamidis Free Acid 12.2 mg Oral Tablet (Fed) (N=21)
Headache (Nervous system disorders) | 4 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT05498701/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT05498701/SAP_001.pdf